CLINICAL TRIAL: NCT03712735
Title: Effect of Programmed Intermittent Epidural Bolus Delivery Rate on the Quality of Labour Analgesia: A Randomized Clinical Trial
Brief Title: Programmed Intermittent Epidural Bolus For Laboring Obstetrical Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H18-02318
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Labor Pain
Keywords: Labor analgesia; Programmed intermittent epidural bolus
MeSH Terms: conditions — Labor Pain | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Bupivacaine 0.08% - fentanyl 2mcg on the following pump settings:
  PIEB flow rate = high; interval = 60 min
  Interventions: Drug: Bupivacaine 0.08% - fentanyl 2mcg
- Group B (Experimental): Bupivacaine 0.08% - fentanyl 2mcg on the following pump settin PIEB flow rate = high; interval = 45 min
  Interventions: Drug: Bupivacaine 0.08% - fentanyl 2mcg
- Group C (Experimental): Bupivacaine 0.08% - fentanyl 2mcg on the following pump settin PIEB flow rate = low; interval = 45 min
  Interventions: Drug: Bupivacaine 0.08% - fentanyl 2mcg

INTERVENTIONS:
Drug: Bupivacaine 0.08% - fentanyl 2mcg — In each arm, bupivacaine and fentanyl are being delivered at different intervals and rates for the maintenance of labor analgesia.

SUMMARY:
Comparison of three programmed intermittent epidural bolus (PIEB) pump settings for maintenance of labour analgesia.

DETAILED DESCRIPTION:
The optimal PIEB and patient controlled epidural administered (PCEA) bolus settings are still unknown. Therefore, in this study, the investigators aim to compare analgesia outcomes both high and low PIEB flow rate settings.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, vertex presentations at term (37-42 weeks gestational age)
* </= 5cm cervical dilation at the time of epidural anesthesia request
* ASA 2-3 patients aged 19 or over who are able to provide informed consent

Exclusion Criteria:

* Contraindications to neuraxial analgesia or risk factors likely to affect placement or function of the epidural
* History of hypersensitivity or idiosyncratic reaction to local anesthetics or opioids
* Current or historical evidence of any significant medical conditions
* Clinical settings in which continuous epidural infusion may be preferable
* Risk factors significantly increasing the need for Cesarean delivery
* Anticipated fetal abnormalities

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Breakthrough pain | Duration of labor with epidural
  Proportion of patients in each group who required a provider administered supplemental bolus for breakthrough pain

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD MMSc, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No